CLINICAL TRIAL: NCT03578445
Title: Utility of EUS-guided Microbiopsies Combined With Auxiliary Molecular Techniques in the Workup of Pancreatic Cystic Lesions
Brief Title: Utility of EUS-guided Microbiopsies in Pancreatic Cystic Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Bojan Kovacevic, Principal Investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-17031060
Record Dates: First submitted 2018-05-28; First posted 2018-07-06 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Pancreatic Cyst; IPMN; Mucinous Cyst; Pancreatic Adenocarcinoma
Keywords: EUS; EUS-FNA; microbiopsy
MeSH Terms: conditions — Pancreatic Cyst; Mucocele

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a pancreatic cystic lesion (Experimental)
  Interventions: Device: EUS-guided microbiopsy; Diagnostic Test: Next Generation Sequencing

INTERVENTIONS:
Device: EUS-guided microbiopsy — Use of EUS-guided through-the-needle microbiopsy forceps for obtainment of tissue from the wall of the cystic lesion
  Other Names: Moray
Diagnostic Test: Next Generation Sequencing — Prevalence of genetic mutations in known cancer-associated genes in the microbiopsy tissue examined using the Ion AmpliSeq Cancer Hotspot Panel v2 (Life Technologies, Carlsbad, USA). The multigene panel explores selected regions of 50 cancer-associated genes, among others KRAS, GNAS, CDKN2A and SMAD4 genes.
  Other Names: NGS

SUMMARY:
The purpose of this study is to determine clinical impact of EUS-guided microbiopsy procedure and supplementary molecular analyses compared to standard diagnostic workup of pancreatic cysts. The hypothesis is that a combination of previously mentioned modalities may change the management of some pancreatic cystic lesions, increase the diagnostic accuracy and optimize the discrimination between high- and low-risk pancreatic cysts.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC) accounts for 6% of all cancer related deaths in Denmark, and the 5-year survival rate is only 8%. PDAC develops from precursor lesions with pancreatic intraepithelial neoplasia (panIN) being the most common, and cystic lesions as a second precursor. Unlike panINs, which are too small for detection with current imaging modalities, cystic lesions of the pancreas are increasingly diagnosed due to the extended use of cross-sectional imaging. Pancreatic cystic lesions may be observed in up to 13.5% of all MRI scans and 3% of all CT scans. There are several types of pancreatic cysts and each of them requires individual management, ranging from no treatment over watchful waiting to surgical resection according to their malignant potential.

Standard diagnostic workup includes cross-sectional imaging of the cystic lesions and, in selected cases endoscopic ultrasound (EUS) with aspiration of cyst fluid by fine needle aspiration (FNA), followed by cyst fluid cytology and tumor marker analysis. The diagnostic algorithm is based on International consensus guidelines established in 2006, and revised in 2012 and 2017, integrating clinical features with EUS-findings. The level of evidence in these guidelines is unfortunately low. A recent meta-analysis concluded that EUS and cyst fluid cytology have low sensitivity (54-63%), whereas the specificity is acceptable (88-92%) for detection of mucinous cysts. Low sensitivity is mainly due to absence of sufficient cellular material in the cyst fluid for definite diagnosis. Tumor marker analysis of cyst fluid, such as carcinoembryonic antigen (CEA), CA 72.4, CA 125, CA 19.9, and CA 15.3, have been studied extensively with CEA being the most accurate marker. A cut-off value of 192 ng/mL for CEA distinguishes mucinous from non-mucinous cysts with a good, albeit imperfect, accuracy of 80%. However, the value will not differentiate between IPMN and MCN, and more importantly, it does not correlate with the level of dysplasia or malignancy.

EUS-guided through-the-needle microbiopsy using the Moray™ forceps is a novel adjunctive. The device can be inserted through a EUS-FNA needle and used to obtain microbiopsies from different tissues in relationship to the gastrointestinal system. This instrument can be used in combination with EUS-FNA to subsequently obtain microbiopsies from the pancreatic cyst wall. Microbiopsies seem to represent a break-through in pre-operative classification of pancreatic cysts, as they provide histological material for examination of tissue architecture not readily accessible in FNA material. However, very little experience has been obtained hitherto. Even though this technique is currently described only in a few studies, it seems feasible and theoretically offers a higher quality of material than what can be obtained by EUS-FNA alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or above
* Able to provide informed consent
* Pancreatic cyst with a diameter of 15 mm or above OR pancreatic cyst of any size with any one of either high-risk stigmata or worrisome features (obstructive jaundice in patients with a cyst in the head of the pancreas, solid component/mural nodule, thickened/enhancing cyst wall, main pancreatic duct ≥ 10 mm or abrupt change of main pancreatic duct diameter with distal atrophy)

Exclusion Criteria:

* Lactating and pregnant females
* Cystic lesions with a predominantly solid component, suspected of malignancy
* Patients with uncorrected coagulopathy (international normalized ratio > 1.5 or platelet count < 50 109/L)
* Patients with previous history of pancreatic cancer
* Patients with a history of major stomach surgery (e.g. Billroth 1 and 2, gastrectomy, gastric bypass, esophagectomy, resection of the liver or pancreas)
* Patients with disseminated malignant disease
* Patients unfit for surgery
* Patients where EUS-guided puncture of the lesion is not presumed technically feasible and/or safe
* Patients with systemic immunosuppressive disease or receiving systemic immunosuppressive treatment
* Patients with a history of recent pancreatitis (within 3 months)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Clinical impact of EUS-guided microbiopsies in patients with pancreatic cystic lesions | 3 weeks
  All patients are evaluated at a multidisciplinary conference prior to microbiopsy procedure. A primary decision is made based on available imaging modalities and/or cyst fluid analysis (operation, follow-up or discontinuation from follow-up). Subsequently, each patient is once again evaluated at a multidisciplinary conference, and a possible change in management is noted. Clinical impact is defined as a proportion of the patients where a change in clinical management is observed.

SECONDARY OUTCOMES:
Technical success of EUS-guided microbiopsy procedure | 3 weeks
  Technical success is defined as a proportion of patients where a pancreatic cystic lesion is successfully punctured by a 19G FNA needle, and where at least one microbiopsy is obtained with the microbiopsy forceps.
Adverse events following EUS-guided microbiopsy procedure | 3 weeks
  Adverse events are defined in concordance with ASGE guidelines (Cotton PB, Eisen GM, Aabakken L et al. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc 2010; 71: 446-454). All patients are contacted by telephone on day 3 following the procedure. Adverse event rate is an overall proportion of the patients where an adverse event is observed.
Diagnostic yield of EUS-guided microbiopsies | 3 weeks
  Diagnostic yield is defined as a proportion of the patients included where a definite histopathological diagnosis could be made on microbiopsy material.
Diagnostic performance of EUS-guided microbiopsies in the surgical subcohort | 2 years
  Sensitivity, specificity as well as positive and negative predictive values are calculated by comparing microbiopsy diagnosis with gold standard (resected specimens).
Diagnostic values of gene mutations (NGS analyses) in microbiopsy material in the surgical subcohort | 2 years
  Sensitivity, specificity as well as positive and negative predictive values are calculated by correlating different mutations with final diagnosis in patients that undergo surgery. NGS analysis is performed using the Ion AmpliSeq Cancer Hotspot Panel v2 (Life Technologies, Carlsbad, USA). The multigene panel explores selected regions of 50 cancer-associated genes, among others KRAS, GNAS, CDKN2A and SMAD4 genes.

CONTACTS AND LOCATIONS:
Locations (1):
- Gastro Unit, Division of Endoscopy, Herlev, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rift CV, Melchior LC, Kovacevic B, Klausen P, Toxvaerd A, Grossjohann H, Karstensen JG, Brink L, Hassan H, Kalaitzakis E, Storkholm J, Scheie D, Hansen CP, Lund EL, Vilmann P, Hasselby JP. Targeted next-generation sequencing of EUS-guided through-the-needle-biopsy sampling from pancreatic cystic lesions. Gastrointest Endosc. 2023 Jan;97(1):50-58.e4. doi: 10.1016/j.gie.2022.08.008. Epub 2022 Aug 12. PMID 35964683